CLINICAL TRIAL: NCT00175149
Title: The Efficacy of 1,25 Dihydroxycholecalciferol on the Cardiovascular System in Patients With Renal Dysfunction
Brief Title: Active Vitamin D Effect on Left Ventricular Hypertrophy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Per Ivarsen (Other)
Responsible Party: Sponsor-Investigator, Per Ivarsen, Consultant, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EX 0203 DK
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism; Left Ventricular Hypertrophy
Keywords: CKD 3-4
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Hypertrophy, Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Given alfacalcidiol. Dose adjusted after PTH level
  Interventions: Drug: Alfacalcidiol
- 2 (No Intervention): The untreated arm

INTERVENTIONS:
Drug: Alfacalcidiol — Alfacalcidiol are given to patientwith CKD 3-4 and secondary hyperparathyrodism. The PTH level is lowered to normal range. with increasing dose of alfacalcidiol and are followed for 6 month.
  Arms: 1

SUMMARY:
Left ventricular hypertrophy (LVH) predicts mortality at start of dialysis. Prevention of of LVH is important. It is not known whether secondary hyperparathyroidism might induce LVH. In the present study patients are randomised to 1.25 dihydroxycholecalciferol or no treatment to study the effect on LVH.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease (S-creatinin > 150 and < 600 mikroM)
* Secondary hyperparathyroidism (Between 3-8 times the upper limit of our PTH assay)
* Stable blood pressure during the last 6 months (less than (160/95)
* B-hemoglobin > 6 mmol/l
* EKG with sinus rhythm and no sign of Q-wave infarction
* Expected follow up 6 month

Exclusion Criteria:

* Pregnancy
* Kidney transplantation
* Malignant disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The effect of dihydroxycholecalciferol on left ventricular hypertrophy | 6 month

SECONDARY OUTCOMES:
Changes in the activity of the renin-angiotensin system | 6 month
Changes in left ventricular function | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Per Ivarsen, MD, PhD, Principal Investigator — Deparment of Renam Medicine C, Skejby Hospital; Per Ivarsen, MD, PhD, Principal Investigator — Deparment of Renal Medicine C, Skejby Hospital
Locations (1):
- Department of Renal Medicne C, Skejby Hospital, Aarhus, Denmark